CLINICAL TRIAL: NCT01568723
Title: Stem Cells And The Origins Of Barrett's Esophagus:Identification Of Novel Biomarkers And Gene Signatures In Barrett's Esophagus
Brief Title: Betrnet Stem Cells and the Origins of Barrett's Esophagus Project 3 RF Ablation
Acronym: BetrnetRF
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenneth K. Wang, Principal Investigator, Mayo Clinic
Other Study IDs: 11-006510; U54CA163004 (NIH)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus; high grade dysplasia; ablation; radiofrequency ablation; esophageal cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsy samples, serum, plasma, buffycoat, cytology brushings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiofrequency ablation: participants with barrett's esophagus with high grade dysplasia who undergo radiofrequency ablation (RFA)
  Interventions: Genetic: response to therapy

INTERVENTIONS:
Genetic: response to therapy — evaluate specific markers for response to therapy at specific intervals pre and post therapy

SUMMARY:
The purpose of this study is to determine biomarkers which can predict response to ablation therapy in patients with Barretts esophagus.

DETAILED DESCRIPTION:
This Project is designed to identify biologically-based and clinically-useful biomarkers of tissue at risk for neoplastic progression as well as of response to ablation therapy. These results will result in improved risk stratification in BE and better targeting of resources for patients who are candidates for ablative therapy, while simultaneously providing key information regarding the origins of Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's esophagus with high grade dysplasia or intramucosal (early) adenocarcinoma.
* BE length ≥ 2 cm and ≤ 8 cm.
* Able to return every 3 months for one year after ablation

Exclusion Criteria:

* Patients who are unable to be compliant with follow-up endoscopies
* patients who cannot tolerate Proton Pump inhibitors
* pre-existing esophageal strictures
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have biopsy proven Barret's esophgus with evidence of specialized intestinal epithelium with high grade dysplasia or early intramucosal carcinoma (mEAC) on histology (confirmed by two pathologists). Patients must have a BE length ≥ 2 cm and ≤ 8 cm.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Response to therapy | one year post ablation
  evaulation will be made at 3 month intervals for one year post ablation

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Wang, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials